CLINICAL TRIAL: NCT04600518
Title: A Retrospective, Multi-center, Single-blind, Pivotal Trial to Assess Clinical Equivalence With Stage II and III Advanced Gastric Cancer Based on the 6th and 8th of the AJCC
Brief Title: Single Patient Classifier (SPC) Prediction for Stage II and III Advanced Gastric Cancer
Acronym: SPRINT
Status: Completed | Type: Observational
Sponsor: Novomics. Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: NM-CTP-04
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2023-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — FFPE samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- SPRINT cohort: stage II and III advanced gastric cancer patients based on the 6th and 8th of the AJCC
  Interventions: Device: nProfiler I Stomach Cancer Assay Kit

INTERVENTIONS:
Device: nProfiler I Stomach Cancer Assay Kit — nProfiler I Stomach Cancer Assay Kit (Novomics Co., Korea)

SUMMARY:
A retrospective, multi-center, single-blind, pivotal trial to assess clinical equivalence with stage II and III advanced gastric cancer based on the 6th and 8th of the AJCC

DETAILED DESCRIPTION:
The safety and effectiveness of nProfiler® 1 Stomach Cancer Assay have been evaluated with stage II and III advanced gastric cancer patients based on the 6th of the American Joint Committee on Cancer (AJCC) through discovery clinical trial (418 patients) and confirmatory clinical trial (684 patients).

The goal of this study, a retrospective, multi-center, single-blind, pivotal trial, is to assess clinical equivalence with stage II and III advanced gastric cancer based on the 6th and 8th of the AJCC and to evaluate prognostic equivalence between surgery only group and adjuvant chemotherapy group in Low risk group.

The study will follow these procedures; Sample screening, Sample Preparation and Sample Criteria Evaluation, Sample enrollment, nProfiler® 1 Stomach Cancer Assay (gastric cancer prognosis prediction), Prognostic Result Report, and Evaluation of Clinical Performance.

ELIGIBILITY:
Inclusion Criteria:

1. Sample providers criteria

   * Male and female adult patients aged 19 years or over
   * Postoperative patients with gastric cancer invading the submucosal layer and having 3 or more lymph nodes metastasis or who with gastric cancer infiltration of muscularis propria and lymph node metastasis (stage II and III advanced gastric cancer patients, 8th of the AJCC)
   * Patients who have not received neoadjuvant chemotherapy and radiotherapy
   * Patients with pathological record and clinical information after surgery from archived FFPE(formalin-fixed paraffin-embedded) samples between 2005 and 2010
   * Patients who have not been included in discovery clinical trial and confirmatory clinical trial
   * Patients who have undergone a radical gastrectomy and who show no evidence of residual tumors as observed with the unaided eye or through a microscope
2. Sample criteria

   * The FFPE tumor specimens in storage have a tumor amount of at least 20% and therefore can be tested.
   * The quantity (not less than 400ng) and quality (A260/280 of not less than 1.8) of RNA are sufficient for analysis.

Exclusion Criteria:

1. Sample providers criteria

   * Male and female patients aged less than 19 years
   * Postoperative patients with gastric cancer invading the mucosa and submucosal layer and having less than 3 lymph nodes metastasis or who with gastric cancer infiltration of muscularis propria without lymph node metastasis (stage II and III advanced gastric cancer patients, 8th of the AJCC)
   * Patients who have received neoadjuvant chemotherapy or radiotherapy
   * Patients without pathological record and clinical information after surgery from archived FFPE samples between 2005 and 2010
   * Patients who have been included in discovery clinical trial and confirmatory clinical trial
   * Patients with residual tumors after surgery
2. Sample criteria

   * The FFPE tumor specimens in storage have a tumor amount of less than 20% and therefore cannot be tested
   * The quantity and quality of RNA are not sufficient for analysis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 19 years or older patients with stage II, III gastric adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 2047 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2023-06-18 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Differences in prognosis | 5 years after the date of surgery for patients in Low risk group and High risk group
  Differences in prognosis between Low risk group and High risk group (AJCC 8th, Advanced gastric cancer stage II and III)
Comparability of prognostic stratification | 5 years after the date of surgery for patients in Low risk group and High risk group
  Comparability of prognostic stratification with stage II and III advanced gastric cancer based on the 6th and 8th of the AJCC
Prognostic equivalence | 5 years after the date of surgery for patients in surgery only group and adjuvant chemotherapy group in Low risk group
  Prognostic equivalence between surgery only group and adjuvant chemotherapy group in Low risk group

SECONDARY OUTCOMES:
Multivariate analysis | 5 years after the date of surgery for patients with stage II-III advanced gastric cancer (8th of the AJCC)
  Multivariate analysis with age, sex, TNM stage, adjuvant-chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Young-Woo Kim, MD., Ph.D., Principal Investigator — National Cancer Center
Locations (1):
- Novomics. Co., Ltd., Seoul, South Korea